CLINICAL TRIAL: NCT02558803
Title: HPV Vaccination: Evaluation of Reminder Prompts for Doses 2 & 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenstrief Institute, Inc. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Merck 21
Record Dates: First submitted 2015-09-18; First posted 2015-09-24 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Human Papilloma Virus Infection Type 11; Human Papilloma Virus Infection Type 16; Human Papilloma Virus Infection Type 18; Human Papilloma Virus Infection Type 6; Cervical Cancer; Genital Warts; Oropharyngeal Cancer
Keywords: HPV Vaccinations; Quadrivalent Vaccine
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata; Oropharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): The clinical team will be left to identify the need for a follow-up HPV vaccine through existing mechanisms
- Simple Reminder (Experimental): A simple reminder prompt in which CHICA will provide an immunization reminder to the physician that the child is eligible for the 2nd or 3rd dose of vaccine.
  Interventions: Behavioral: Simple Reminder

INTERVENTIONS:
Behavioral: Simple Reminder — A simple reminder prompt in which CHICA will provide an immunization reminder to the physician that the child is eligible for the 2nd or 3rd dose of vaccine.
  Arms: Simple Reminder

SUMMARY:
Randomized, 2-arm observational study. The 2 arms (randomized at the level of health care provider) will be: 1. usual practice; 2. automated reminders to recommend 2nd and 3rd doses of HPV vaccine for eligible male and female adolescents who have initiated vaccination.

DETAILED DESCRIPTION:
The study team plans to conduct a randomized clinical trial with three arms: (1) usual care, (2) the simple reminder, and (3) the simple reminder plus the script. Randomization will be carried out at the physician level at each clinical site, to ensure that all three treatment arms are represented in each clinic. The primary outcome, HPV vaccine acceptance, will be assessed for each study participant.

This study will be implemented through the Child Health Improvement through Computer Automation system (CHICA). CHICA is a computer based clinical decision support system that has been operating in the Wishard/Eskenazi system since 2004. CHICA now operates in 5 clinics in the health system and has served well over 37,000 children. CHICA supports primary pediatric care, supporting screening, counseling, anticipatory guidance, vaccinations, and chronic disease diagnosis and management.

CHICA is unique in several respects. These include a unique tailored, scannable paper interface, a prioritization scheme that assures the highest priority reminders are given to physicians, and the ability to collect data directly from families in the waiting room. CHICA acts as a front end to the Regenstrief Medical Record System (RMRS), the electronic medical record for the Eskenazi health system. The RMRS and CHICA communicate using industry standard HL7 communication protocols.

When a patient checks into a CHICA clinic, CHICA receives an HL7 ADT (registration) message. In response CHICA requests a download of the patient's record from the RMRS. CHICA applies a set of Arden Syntax rules to the patient's data to select 20 yes/no questions that are printed. The family answers these questions by checking boxes. The nurse or medical assistant enters height, weight, etc. on the same form and the form is scanned. The data enter CHICA's database through optical mark recognition and optical character recognition. Recently we have begun converting from this scannable paper format to electronic tablets.

ELIGIBILITY:
Inclusion Criteria:

Provider Criteria

* All pediatricians and nurse practitioners who provide health care at the 5 CHICA clinics will be included in this study

Subject Criteria

* Patients will be 11-17 year old
* Males and females
* A visit to at least one of the five CHICA clinics
* Eligible for the 2nd or 3rd dose of HPV vaccine

Exclusion Criteria:

* Patients in the eligible age range who have not started or have completed the HPV vaccine series will be excluded

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1305 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rate of physician-targeted automated HPV vaccination reminders on 2nd and 3rd dose HPV vaccination rates among 11-17 year old male and female patients | Six Months
  To evaluate the rate of physician-targeted automated HPV vaccination reminders on 2nd and 3rd dose HPV vaccination rates among 11-17 year old male and female patients who have received 1 or 2 doses of vaccine.

SECONDARY OUTCOMES:
Assessment of Physician Acceptance of the Prompts | Six Months
  The study team will compare changes in vaccination rates with qualitative feedback from providers.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University
Locations (5):
- United States (5):
  - Eskenazi Health Outpatient Care Center, Indianapolis, Indiana
  - Eskenazi Health Center Blackburn, Indianapolis, Indiana
  - Eskenazi Health Center Forest Manor, Indianapolis, Indiana
  - Eskenazi Health West 38th Street, Indianapolis, Indiana
  - Eskenazi Health Center Pecar, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No
Individual provider data will not be made available.

REFERENCES:
- [Background] Parkin DM, Bray F. Chapter 2: The burden of HPV-related cancers. Vaccine. 2006 Aug 31;24 Suppl 3:S3/11-25. doi: 10.1016/j.vaccine.2006.05.111. PMID 16949997
- [Background] Giuliano AR, Anic G, Nyitray AG. Epidemiology and pathology of HPV disease in males. Gynecol Oncol. 2010 May;117(2 Suppl):S15-9. doi: 10.1016/j.ygyno.2010.01.026. Epub 2010 Feb 6. PMID 20138345
- [Background] Chaturvedi AK. Beyond cervical cancer: burden of other HPV-related cancers among men and women. J Adolesc Health. 2010 Apr;46(4 Suppl):S20-6. doi: 10.1016/j.jadohealth.2010.01.016. PMID 20307840
- [Background] Haupt RM, Sings HL. The efficacy and safety of the quadrivalent human papillomavirus 6/11/16/18 vaccine gardasil. J Adolesc Health. 2011 Nov;49(5):467-75. doi: 10.1016/j.jadohealth.2011.07.003. Epub 2011 Sep 9. PMID 22018560
- [Background] Arnheim-Dahlstrom L, Pasternak B, Svanstrom H, Sparen P, Hviid A. Autoimmune, neurological, and venous thromboembolic adverse events after immunisation of adolescent girls with quadrivalent human papillomavirus vaccine in Denmark and Sweden: cohort study. BMJ. 2013 Oct 9;347:f5906. doi: 10.1136/bmj.f5906. PMID 24108159
- [Background] Scheller NM, Svanstrom H, Pasternak B, Arnheim-Dahlstrom L, Sundstrom K, Fink K, Hviid A. Quadrivalent HPV vaccination and risk of multiple sclerosis and other demyelinating diseases of the central nervous system. JAMA. 2015 Jan 6;313(1):54-61. doi: 10.1001/jama.2014.16946. PMID 25562266
- [Background] Ojha RP, Jackson BE, Tota JE, Offutt-Powell TN, Singh KP, Bae S. Guillain-Barre syndrome following quadrivalent human papillomavirus vaccination among vaccine-eligible individuals in the United States. Hum Vaccin Immunother. 2014;10(1):232-7. doi: 10.4161/hv.26292. Epub 2013 Sep 6. PMID 24013368
- [Background] Klein NP, Hansen J, Chao C, Velicer C, Emery M, Slezak J, Lewis N, Deosaransingh K, Sy L, Ackerson B, Cheetham TC, Liaw KL, Takhar H, Jacobsen SJ. Safety of quadrivalent human papillomavirus vaccine administered routinely to females. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1140-8. doi: 10.1001/archpediatrics.2012.1451. PMID 23027469
- [Background] Pedersen C, Petaja T, Strauss G, Rumke HC, Poder A, Richardus JH, Spiessens B, Descamps D, Hardt K, Lehtinen M, Dubin G; HPV Vaccine Adolescent Study Investigators Network. Immunization of early adolescent females with human papillomavirus type 16 and 18 L1 virus-like particle vaccine containing AS04 adjuvant. J Adolesc Health. 2007 Jun;40(6):564-71. doi: 10.1016/j.jadohealth.2007.02.015. PMID 17531764
- [Background] Reisinger KS, Block SL, Lazcano-Ponce E, Samakoses R, Esser MT, Erick J, Puchalski D, Giacoletti KE, Sings HL, Lukac S, Alvarez FB, Barr E. Safety and persistent immunogenicity of a quadrivalent human papillomavirus types 6, 11, 16, 18 L1 virus-like particle vaccine in preadolescents and adolescents: a randomized controlled trial. Pediatr Infect Dis J. 2007 Mar;26(3):201-9. doi: 10.1097/01.inf.0000253970.29190.5a. PMID 17484215
- [Background] Baandrup L, Blomberg M, Dehlendorff C, Sand C, Andersen KK, Kjaer SK. Significant decrease in the incidence of genital warts in young Danish women after implementation of a national human papillomavirus vaccination program. Sex Transm Dis. 2013 Feb;40(2):130-5. doi: 10.1097/OLQ.0b013e31827bd66b. PMID 23324976
- [Background] Ali H, Donovan B, Wand H, Read TR, Regan DG, Grulich AE, Fairley CK, Guy RJ. Genital warts in young Australians five years into national human papillomavirus vaccination programme: national surveillance data. BMJ. 2013 Apr 18;346:f2032. doi: 10.1136/bmj.f2032. PMID 23599298
- [Background] Ali H, Guy RJ, Wand H, Read TR, Regan DG, Grulich AE, Fairley CK, Donovan B. Decline in in-patient treatments of genital warts among young Australians following the national HPV vaccination program. BMC Infect Dis. 2013 Mar 18;13:140. doi: 10.1186/1471-2334-13-140. PMID 23506489
- [Background] Elam-Evans LD, Yankey D, Jeyarajah J, Singleton JA, Curtis RC, MacNeil J, Hariri S; Immunization Services Division, National Center for Immunization and Respiratory Diseases; Centers for Disease Control and Prevention (CDC). National, regional, state, and selected local area vaccination coverage among adolescents aged 13-17 years--United States, 2013. MMWR Morb Mortal Wkly Rep. 2014 Jul 25;63(29):625-33. PMID 25055186
- [Background] Brewer NT, Gottlieb SL, Reiter PL, McRee AL, Liddon N, Markowitz L, Smith JS. Longitudinal predictors of human papillomavirus vaccine initiation among adolescent girls in a high-risk geographic area. Sex Transm Dis. 2011 Mar;38(3):197-204. doi: 10.1097/OLQ.0b013e3181f12dbf. PMID 20838362
- [Background] Guerry SL, De Rosa CJ, Markowitz LE, Walker S, Liddon N, Kerndt PR, Gottlieb SL. Human papillomavirus vaccine initiation among adolescent girls in high-risk communities. Vaccine. 2011 Mar 9;29(12):2235-41. doi: 10.1016/j.vaccine.2011.01.052. Epub 2011 Feb 1. PMID 21288799
- [Background] Donahue KL, Stupiansky NW, Alexander AB, Zimet GD. Acceptability of the human papillomavirus vaccine and reasons for non-vaccination among parents of adolescent sons. Vaccine. 2014 Jun 30;32(31):3883-5. doi: 10.1016/j.vaccine.2014.05.035. Epub 2014 May 18. PMID 24844150
- [Background] Kester LM, Zimet GD, Fortenberry JD, Kahn JA, Shew ML. A national study of HPV vaccination of adolescent girls: rates, predictors, and reasons for non-vaccination. Matern Child Health J. 2013 Jul;17(5):879-85. doi: 10.1007/s10995-012-1066-z. PMID 22729660
- [Background] Vadaparampil ST, Kahn JA, Salmon D, Lee JH, Quinn GP, Roetzheim R, Bruder K, Malo TL, Proveaux T, Zhao X, Halsey N, Giuliano AR. Missed clinical opportunities: provider recommendations for HPV vaccination for 11-12 year old girls are limited. Vaccine. 2011 Nov 3;29(47):8634-41. doi: 10.1016/j.vaccine.2011.09.006. Epub 2011 Sep 14. PMID 21924315
- [Background] Evans, G. and A. Bostrom, The evolution of vaccine risk communication in the United States: 1982-2002, in Jordan report 20th anniversary: Accelerated development of vaccines 2002, A. National Institute of and D. Infectious, Editors. 2002, U.S. Department of Health and Human Services, National Institute of Allergy and Infectious Diseases: Washington, D.C. p. 58-71.
- [Background] Esposito S, Bosis S, Pelucchi C, Begliatti E, Rognoni A, Bellasio M, Tel F, Consolo S, Principi N. Pediatrician knowledge and attitudes regarding human papillomavirus disease and its prevention. Vaccine. 2007 Aug 29;25(35):6437-46. doi: 10.1016/j.vaccine.2007.06.053. Epub 2007 Jul 16. PMID 17673339
- [Background] Schnatz PF, Humphrey K, O'Sullivan DM. Assessment of the perceptions and administration of the human papillomavirus vaccine. J Low Genit Tract Dis. 2010 Apr;14(2):103-7. doi: 10.1097/LGT.0b013e3181b240ca. PMID 20354417
- [Background] Kahn JA. Vaccination as a prevention strategy for human papillomavirus-related diseases. J Adolesc Health. 2005 Dec;37(6 Suppl):S10-6. doi: 10.1016/j.jadohealth.2005.08.018. PMID 16310136
- [Background] Ko EM, Missmer S, Johnson NR. Physician attitudes and practice toward human papillomavirus vaccination. J Low Genit Tract Dis. 2010 Oct;14(4):339-45. doi: 10.1097/LGT.0b013e3181dca59c. PMID 20885162
- [Background] Carroll AE, Bauer NS, Dugan TM, Anand V, Saha C, Downs SM. Use of a computerized decision aid for ADHD diagnosis: a randomized controlled trial. Pediatrics. 2013 Sep;132(3):e623-9. doi: 10.1542/peds.2013-0933. Epub 2013 Aug 19. PMID 23958768
- [Background] Carroll AE, Biondich P, Anand V, Dugan TM, Downs SM. A randomized controlled trial of screening for maternal depression with a clinical decision support system. J Am Med Inform Assoc. 2013 Mar-Apr;20(2):311-6. doi: 10.1136/amiajnl-2011-000682. Epub 2012 Jun 28. PMID 22744960
- [Background] Carroll AE, Biondich PG, Anand V, Dugan TM, Sheley ME, Xu SZ, Downs SM. Targeted screening for pediatric conditions with the CHICA system. J Am Med Inform Assoc. 2011 Jul-Aug;18(4):485-90. doi: 10.1136/amiajnl-2011-000088. PMID 21672910
- [Background] Fu LY, Bonhomme LA, Cooper SC, Joseph JG, Zimet GD. Educational interventions to increase HPV vaccination acceptance: a systematic review. Vaccine. 2014 Apr 7;32(17):1901-20. doi: 10.1016/j.vaccine.2014.01.091. Epub 2014 Feb 14. PMID 24530401
- [Background] Mayne SL, duRivage NE, Feemster KA, Localio AR, Grundmeier RW, Fiks AG. Effect of decision support on missed opportunities for human papillomavirus vaccination. Am J Prev Med. 2014 Dec;47(6):734-44. doi: 10.1016/j.amepre.2014.08.010. Epub 2014 Nov 18. PMID 25455116
- [Background] Fiks AG, Grundmeier RW, Mayne S, Song L, Feemster K, Karavite D, Hughes CC, Massey J, Keren R, Bell LM, Wasserman R, Localio AR. Effectiveness of decision support for families, clinicians, or both on HPV vaccine receipt. Pediatrics. 2013 Jun;131(6):1114-24. doi: 10.1542/peds.2012-3122. Epub 2013 May 6. PMID 23650297
- [Background] Perkins RB, Zisblatt L, Legler A, Trucks E, Hanchate A, Gorin SS. Effectiveness of a provider-focused intervention to improve HPV vaccination rates in boys and girls. Vaccine. 2015 Feb 25;33(9):1223-9. doi: 10.1016/j.vaccine.2014.11.021. Epub 2014 Nov 24. PMID 25448095
- [Background] Markowitz LE, Hariri S, Lin C, Dunne EF, Steinau M, McQuillan G, Unger ER. Reduction in human papillomavirus (HPV) prevalence among young women following HPV vaccine introduction in the United States, National Health and Nutrition Examination Surveys, 2003-2010. J Infect Dis. 2013 Aug 1;208(3):385-93. doi: 10.1093/infdis/jit192. Epub 2013 Jun 19. PMID 23785124
- [Background] Zimet GD, Rosberger Z, Fisher WA, Perez S, Stupiansky NW. Beliefs, behaviors and HPV vaccine: correcting the myths and the misinformation. Prev Med. 2013 Nov;57(5):414-8. doi: 10.1016/j.ypmed.2013.05.013. Epub 2013 May 31. PMID 23732252
- [Background] Shojania KG, Jennings A, Mayhew A, Ramsay CR, Eccles MP, Grimshaw J. The effects of on-screen, point of care computer reminders on processes and outcomes of care. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD001096. doi: 10.1002/14651858.CD001096.pub2. PMID 19588323
- [Background] Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. Milbank Q. 2004;82(4):581-629. doi: 10.1111/j.0887-378X.2004.00325.x. PMID 15595944
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Anand V, Biondich PG, Liu G, Rosenman M, Downs SM. Child Health Improvement through Computer Automation: the CHICA system. Stud Health Technol Inform. 2004;107(Pt 1):187-91. PMID 15360800
- [Background] Anand V, Carroll AE, Downs SM. Automated primary care screening in pediatric waiting rooms. Pediatrics. 2012 May;129(5):e1275-81. doi: 10.1542/peds.2011-2875. Epub 2012 Apr 16. PMID 22508925
- [Background] Biondich PG, Downs SM, Anand V, Carroll AE. Automating the recognition and prioritization of needed preventive services: early results from the CHICA system. AMIA Annu Symp Proc. 2005;2005:51-5. PMID 16779000
- [Background] Downs SM, Uner H. Expected value prioritization of prompts and reminders. Proc AMIA Symp. 2002:215-9. PMID 12463818
- [Background] Downs SM, Zhu V, Anand V, Biondich PG, Carroll AE. The CHICA smoking cessation system. AMIA Annu Symp Proc. 2008 Nov 6;2008:166-70. PMID 18998823
- [Background] Bauer, N.S., et al., Computer Decision Support to Improve Autism Screening and Care in Community Pediatric Clinics. Infants & Young Children, 2013. 26(4): p. 306-317.
- [Background] Denzin, N.K. and Y.S. Lincoln, The Sage handbook of qualitative research. Vol. 4th. 2011, Thousand Oaks, CA: Sage.
- [Background] Braun, V. and V. Clarke, Using thematic analysis in psychology. Qualitative Research in Psychology, 2006. 3: p. 77-101.
- [Background] Fleiss JL, Tytun A, Ury HK. A simple approximation for calculating sample sizes for comparing independent proportions. Biometrics. 1980 Jun;36(2):343-6. PMID 26625475
- [Derived] Wilkinson TA, Dixon BE, Xiao S, Tu W, Lindsay B, Sheley M, Dugan T, Church A, Downs SM, Zimet G. Physician clinical decision support system prompts and administration of subsequent doses of HPV vaccine: A randomized clinical trial. Vaccine. 2019 Jul 18;37(31):4414-4418. doi: 10.1016/j.vaccine.2019.05.004. Epub 2019 Jun 11. PMID 31201057